CLINICAL TRIAL: NCT01735669
Title: Open Randomized Controlled Trial to Evaluate the Efficacy and Safety of Remifentanil Versus Nitrous Oxide in External Cephalic Version at Term in Singleton Pregnancy in Breech Presentation
Acronym: REMIVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Cruces (Other)
Responsible Party: Principal Investigator, Jorge Burgos, PROFESSOR, Hospital de Cruces
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIVER
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Non-cephalic Presentation; Inhalation of Nitrous Oxide; Pregnancy Complications; Complications; Cesarean Section; Fetus or Neonate Affected by External Version Before Labor
Keywords: Remifentanil; Breech presentation; Nitrous oxide; Pregnancy complications; Caesarean section; Fetal version
MeSH Terms: conditions — Pregnancy Complications; Breech Presentation | interventions — Remifentanil; Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental): External cephalic version at term under Remifentanil perfusion
  Interventions: Drug: Remifentanil
- Nitrous oxide (Active Comparator): External cephalic version at term under Nitrous oxide inhalation
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Remifentanil
  Other Names: CAS- NUMBER: 132875-61-7
  Arms: Remifentanil
Drug: Nitrous Oxide
  Other Names: CAS_NUMBER:10024-97-2
  Arms: Nitrous oxide

SUMMARY:
Objectives: The objective is to demonstrate the superiority of remifentanil versus nitrous oxide as adjuvant analgesic treatment to increase the chances of success of external cephalic version in the management of non-cephalic presentation in women with singleton pregnancy at term. Another objective is to compare their safety, tolerability and acceptability.

Methodology: single-center clinical trial, randomized, open, parallel-group and sequential design, with active comparator. Pragmatic approach. Sequential design of O'Brien-Fleming with two interim analysis. Analysis by intention to treat. Comparison of the rate of successful version, referred to analgesic effect, safety, caesarean rates and acceptability rate of the procedure for pregnant women.

DETAILED DESCRIPTION:
External cephalic version is a procedure with clear benefits, but its realization is painful for the patient. Studies have shown that this pain limits external cephalic version efforts and therefore it negatively influences its success rate. In addition, any painful procedure has worse acceptance by patients so that its implementation is slow and not always universal. In this context, measures to reduce this pain could improve the success rate and acceptance of the procedure. All studies that have focused on reducing pain in external cephalic version have been made with regional anaesthetic techniques, epidural or spinal analgesia. Given the heterogeneity and the small number of studies there is still no conclusive data to make recommendations for regional anaesthesia in the external cephalic version. The introduction of regional anaesthesia can bring benefits to the version but it is not without drawbacks. This is an invasive anaesthetic technique that can reduce the security of the procedure and lead to longer hospital stay for the patient by the blockade that produces in the lower extremities. This in turn is associated with increased discomfort and costs of the procedure.

Cruces University Hospital has wide experience in carrying out external cephalic version procedures, being one of Spanish leading hospitals in terms of number of procedures and success rate. Currently external cephalic version procedures include analgesic support using nitrous oxide due to the combination of moderate analgesic activity and substantial ease of use.

The investigators belief is that the use of an opioid with advantageous pharmacokinetic properties and powerful analgesic effect as an adjunctive therapy during the course of external cephalic version procedures may become an efficacious and safe alternative, leading to increased pain relief and improved external cephalic version success rates. Its use requires, however, specific personnel and organizational facilities such as access to anesthetic support that can impede its widespread use. Therefore, the investigators is committed to explore feasibility and practical implementation factors as well as comparative efficacy and safety of this approach in non-cephalic presentation.

The investigators conducted a study to evaluate the effect of nitrous oxide as an adjunctive to external cephalic version and we observed a slight decrease in patient reported pain (visual analogous scale), with no effect on the rate of success. Currently, in the protocol of Cruces University Hospital the administration of nitrous oxide during the manoeuvres of the external cephalic version is routine practice. The investigators consider that the analgesic remifentanil is a better option for the external cephalic version than nitrous oxide by the combination of rapid onset of effect, with analgesic potency similar to regional anaesthesia and rapid metabolism that prevents their accumulation in tissues.

The lack of existing evidence on this issue, hence, prompts the investigators to conduct this pilot clinical trial aimed to assess scientific as well as logistical aspects involved in the performance of external cephalic version in non-cephalic presentation.

ELIGIBILITY:
Inclusion Criteria:

1. pregnancy at term (≥ 37 weeks)
2. singleton foetus in non-cephalic presentation
3. correct foetal cardiotocographic record
4. obstetrical ultrasound examination without findings of serious foetal malformations
5. indication for the performance of ECV
6. acceptance of ECV
7. age ≥ 18 years
8. signature of informed consent

Exclusion Criteria:

1. previous version in the same pregnancy (previous ECV in a different pregnancy allowed)
2. contraindications to ECV: 1-placenta praevia, 2- placental abruption, 3-oligohydramnios (SPD <2), 4-foetal compromise 5-foetal death, 6-severe malformations, 7-multiple pregnancy, 8- Rh sensitization, 9- uterine abnormalities, 10- clotting disorders;
3. contraindications to Nitrous Oxide: 1-patients who require pure oxygen ventilation 2- intracranial hypertension 3- disorders of consciousness that impede the cooperation of the patient, 4-pneumothorax; 5-emphysematous bulla, 6-pulmonary embolism; 7-immersion accident, 8-bloating abdominal trauma 9- facial trauma that affects the area of application of the mask,10- patients who received the type gases SF6, C3F8, C2F6 (used in eye surgery), at least in the previous three months.
4. contraindications for remifentanil: hypersensitivity to remifentanil, fentanyl or fentanyl analogs or to any component of its formulation (according to technical requirements by manufacturer).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Success rate of ECV in singleton pregnancies in breech presentation at term | 5 minutes

SECONDARY OUTCOMES:
Rate of adverse events and severity | 30 days
  Metrics (analysis)
Pain Scores on the Visual Analog Scale | 60 min
  Metrics (scale)
Rate of non-cephalic presentation in the delivery | 30 days
  Metrics (analysis)
Caesarean rate | 30 days
  Metrics (analysis)
Rate of women who would recommend the procedure | 60 min
  Metrics (questionnaire)
Rate of women who would repeat the procedure | 60 min
  Metrics (questionnaire)
Influence of the analgesia in the rate of women who would repeat the procedure | 60 min
  Metrics (questionnaire)
Influence of the analgesia in the rate of women who would recommend the procedure | 60 min
  Metrics (questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Cruces, Barakaldo, Bizkaia, Spain